CLINICAL TRIAL: NCT00360737
Title: Pharmacokinetics of a Heptavalent Equine-derived Botulinum Antitoxin (NP-018)
Brief Title: Safety Study of 7 Botulinum Antitoxin Serotypes Derived From Horses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AA24424 BT-001
Record Dates: First submitted 2006-07-19; First posted 2006-08-07 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Clinical Trials; Investigational Drug; Healthy Volunteers; Botulinum Antitoxin; Phoenix, Arizona
MeSH Terms: interventions — Botulinum Antitoxin

STUDY DESIGN:
Intervention Model Description: 40 subjects will receive 1 or 2 vials of NP-018 intravenously. 20 subjects will be randomized into each arm of the study.
Who Masked: Participant, Investigator
Masking Description: In order to maintain the blind of the study, equivalent volumes will be administered to each subject. Each subject will receive 1 infusion consisting of 2 bags. Subjects randomized to receive 2 vials of NP 018 will be administered approximately 224 mL of NP 018 in saline while subjects receiving 1 vial of NP 018 will be administered approximately 112 mL of NP 018 in saline followed by 112 mL of 0.9% saline. This will ensure the blind is maintained, as equivalent volumes will be administered and the rate of protein administration will be equivalent during the first 112 mL of fluid infused.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NP-018 - 1 vial (Experimental): Subjects received one vials of NP-018 administered intravenously.
  Interventions: Biological: Botulinum Antitoxin Heptavalent (A B C D E F G) - (EQUINE)
- NP-018 - 2 vials (Experimental): Subjects receive two vials of NP-018 administered intravenously.
  Interventions: Biological: Botulinum Antitoxin Heptavalent (A B C D E F G) - (EQUINE)

INTERVENTIONS:
Biological: Botulinum Antitoxin Heptavalent (A B C D E F G) - (EQUINE) — Biological/Vaccine NP-018 (heptavalent equine-derived botulinum antitoxin) is prepared from pooled plasma obtained from horses that have been immunized against one of seven botulinum antitoxins (A-G). .
  Other Names: Botulism Antitoxin (BAT)

SUMMARY:
The primary purpose of the study is to evaluate the safety of the 7 Botulinum Antitoxin Serotypes derived from horses using various laboratory measurements, clinical examinations and adverse events. In addition, following intravenous (injected into the vein) administration assessing how much 7 Botulinum Antitoxin remains in the body.

DETAILED DESCRIPTION:
Clostridial toxins are amongst the most toxic substances known to science (Middlebrook, 1995). In the United States and other countries, human exposure to Clostridium botulinum toxins usually occurs through food poisoning, wound botulism and colonizing infections in neonates. Recent events have heightened concern about the possibility of botulinum toxins being used in a bioterrorist attack. In order to be prepared for a biological attack as well as the usual human exposures, numerous therapeutic products have been or currently are undergoing development to treat or prevent botulism, including the use of human or equine derived antibodies for post-exposure prophylaxis of botulinum toxin exposure (Gelzleichter et al, 1999; Hibbs et al, 1996; Metzger and Lewis, 1979 and Keller and Stiehm, 2000).

Botulinum antitoxins have been in use to treat adult exposure to botulinum toxin for at least 40 years (Cupo et al, 2001). The use of botulinum antitoxins to treat individuals exposed to botulinum toxin is similar to the use of passive immune therapy with immune globulins collected from immunized or convalescing human donors to treat a wide range of bacterial and viral infectious diseases (Chippaux et al, 1998).

NP-018 (heptavalent equine-derived botulinum antitoxin) is prepared from plasma obtained from horses that have been immunized with a specific subtype of botulinum toxoid and toxin. Each individual horse is immunized against a single botulinum toxin subtype. Plasma is pooled from horses that have been immunized with the same botulinum toxin subtype. For each antitoxin serotype (A-G), a despeciated product will be produced by pepsin digestion of the IgG monomer in the equine plasma, yielding predominantly F(ab¢)2 fragment. Following the formulation, the seven antitoxin serotypes will be blended into a heptavalent product and filled into single-use vials.

The present clinical study is intended to assess the pharmacokinetics and safety of NP 018 following intravenous administration. The pharmacokinetics of NP 018 will be comparable to other equine derived antitoxin products. NP 018 will be safe to administer to normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index of 20 to 30 with minimum body weight of 111 lb (50 kg).
* For female subjects that are not surgically sterilized, willingness to use an effective method of contraception throughout the trial including:
* Using hormonal contraception (oral or injectable or implant) continuously for 3 months prior to the start of the trial and willing to continue to use hormonal contraception throughout the entire trial.
* IUD inserted at least 2 months prior to dosing.
* For female subjects who are postmenopausal less than 2 years an FSH >= 40 mIU/mL must be obtained. IF the FSH is < 40 mIU/mL the subject must agree to use an acceptable form of contraception (see above for acceptable forms of contraception.
* Normal and healthy as determined by medical history, physical examination, ECG, vital signs and test of liver, kidney and hematological functions.
* Written Informed Consent

Exclusion Criteria:

* Any known or documented allergies to horses (e.g. rash, wheezing, rhinitis etc. after exposure to horses)
* Any known or documented allergies to horse serum (observation of adverse events after treatment with any kind of products containing horse serum)
* Any severe food allergies, seasonal allergies or hay fever requiring therapy such as treatment with immunosuppressive drugs
* Known acute or chronic asthma requiring treatment with immunosuppressive drugs
* History of hypersensitivity to blood products derived from a human or equine source
* Heavy smokers (>10 cigarettes a day)
* Use of nicotine containing products
* Use of any investigational product within the past 30 days
* Pregnancy or lactation
* Positive serological test for HIV, HBV, or HCV
* History of, or suspected substance abuse problem (including alcohol) or failure of alcohol or drug screen at screening or at baseline
* Individuals with a history of allergy to latex or rubber
* Hemoglobin level of < 12 g/dL.
* Significant blood loss or blood donation within 56 days prior to dosing.
* Any plasma donation within 7 days prior to dosing.
* Demonstrated potential for allergic reaction to NP-018 based on positive horse dander (E3) IgE test or positive NP-018 skin sensitivity test prior to dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07; Primary Completion 2006-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Subjects with adverse events over the course of the study | From Screening Day 1 to Day 28 or early withdrawal
  Number of subjects with AEs and severity of AEs up to Day 28
Subjects with serious adverse events over the course of the study | From Screening Day 1 to Day 28 or early withdrawal
  Number of subjects with SAEs up to Day 28

SECONDARY OUTCOMES:
PK analysis for all 7 botulinum antitoxins: AUC0-t | Day Screening 2, Day 0 -30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  AUC0-t (area under the serum concentration versus time curve, from time 0 to the last measurable concentration, as calculated by the linear trapezoidal method) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration
PK analysis for all 7 botulinum antitoxins: AUC0-inf | Screening Day 2, Day 0- 30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  AUC0-inf (area under the serum concentration versus time curve from time 0 to infinity) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration
PK analysis for all 7 botulinum antitoxins: AUC0-t/AUC0-inf | Screening Day 2, Day 0- 30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  AUC0-t/AUC0-inf (ratio of AUC0-t to AUC0-inf) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration
PK analysis for all 7 botulinum antitoxins: Cmax | Screening Day 2, Day 0- 30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  Cmax (maximum measured serum concentration over the time span specified) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration
PK analysis for all 7 botulinum antitoxins: Tmax | Screening Day 2, Day 0- 30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  Tmax (time of the maximum measured serum concentration) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration
PK analysis for all 7 botulinum antitoxins: t½ | Screening Day 2, Day 0- 30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  t½ (apparent first-order terminal elimination half-life) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration
PK analysis for all 7 botulinum antitoxins: Cl | Screening Day 2, Day 0- 30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  Cl (clearance of NP-018) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration
PK analysis for all 7 botulinum antitoxins: Vd | Screening Day 2, Day 0- 30 minutes, 4 hours, 8 hours, Day 1 [24 hours], Day 3, Day 7, Day 14, Day 21, Day 28 or early withdrawal
  Vd (initial volume of distribution) will be calculated for all 7 botulinum antitoxins for each subject after NP-018 administration

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Allison, M.D., Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States

REFERENCES:
- [Background] Middlebrook JL. Protection strategies against botulinum toxin. Adv Exp Med Biol. 1995;383:93-8. doi: 10.1007/978-1-4615-1891-4_11. No abstract available. PMID 8644518
- [Background] Gelzleichter TR, Myers MA, Menton RG, Niemuth NA, Matthews MC, Langford MJ. Protection against botulinum toxins provided by passive immunization with botulinum human immune globulin: evaluation using an inhalation model. J Appl Toxicol. 1999 Dec;19 Suppl 1:S35-8. doi: 10.1002/(sici)1099-1263(199912)19:1+3.0.co;2-9. PMID 10594898
- [Background] Hibbs RG, Weber JT, Corwin A, Allos BM, Abd el Rehim MS, Sharkawy SE, Sarn JE, McKee KT Jr. Experience with the use of an investigational F(ab')2 heptavalent botulism immune globulin of equine origin during an outbreak of type E botulism in Egypt. Clin Infect Dis. 1996 Aug;23(2):337-40. doi: 10.1093/clinids/23.2.337. PMID 8842274
- [Background] Metzger JF, Lewis GE Jr. Human-derived immune globulins for the treatment of botulism. Rev Infect Dis. 1979 Jul-Aug;1(4):689-92. doi: 10.1093/clinids/1.4.689. PMID 399376
- [Background] Keller MA, Stiehm ER. Passive immunity in prevention and treatment of infectious diseases. Clin Microbiol Rev. 2000 Oct;13(4):602-14. doi: 10.1128/CMR.13.4.602. PMID 11023960
- [Background] Cupo P, de Azevedo-Marques MM, Sarti W, Hering SE. Proposal of abolition of the skin sensitivity test before equine rabies immune globulin application. Rev Inst Med Trop Sao Paulo. 2001 Jan-Feb;43(1):51-3. doi: 10.1590/s0036-46652001000100010. PMID 11246284
- [Background] Chippaux JP, Lang J, Eddine SA, Fagot P, Rage V, Peyrieux JC, Le Mener V. Clinical safety of a polyvalent F(ab')2 equine antivenom in 223 African snake envenomations: a field trial in Cameroon. VAO (Venin Afrique de l'Ouest) Investigators. Trans R Soc Trop Med Hyg. 1998 Nov-Dec;92(6):657-62. doi: 10.1016/s0035-9203(98)90802-1. PMID 10326114